CLINICAL TRIAL: NCT00989404
Title: A Randomized, Placebo Controlled, 3-Way Crossover Study to Investigate the Safety, Tolerability, and Pharmacokinetics of Repeat Dose Zanamivir/Placebo 10mg Administered Twice Daily for 5 Days by a Rotahaler Compared to the Diskhaler in Healthy Subjects
Brief Title: Crossover Study to Investigate the Safety, Tolerability, and Pharmacokinetics of Repeat Dose Zanamivir/Placebo Via Devices Administered Twice Daily for 5 Days
Acronym: NAI113625
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 113625
Record Dates: First submitted 2009-09-24; First posted 2009-10-05 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Influenza A Virus, H1N1 Subtype
Keywords: pk; healthy subjects; influenza virus; Safety; pandemic
MeSH Terms: interventions — Zanamivir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Period (Experimental): 10 mg BID Zanamivir or placebo for 5 days
  Interventions: Drug: Zanamivir

INTERVENTIONS:
Drug: Zanamivir — Rotahaler placebo 10mg BID 5 days
Drug: Zanamivir — Rotahaler Zanamivir 10mg BID 5 days
Drug: Zanamivir — Diskhaler Zanamivir 10mg BID 5 days

SUMMARY:
The purpose of this study is to compare the safety and tolerability of Zanamivir using a Rotahaler device presentation to placebo within the Rotahaler presentation and to the Diskhaler device.

DETAILED DESCRIPTION:
The purpose of this study is to compare the safety and tolerability of Zanamivir using a Rotahaler to placebo within the Rotahaler presentation and to the Diskhaler. Eighteen subjects will receive each of three treatments for 5 days in a 3-way crossover design.

ELIGIBILITY:
Inclusion Criteria:

* The subject is healthy as judged by a responsible physician with no clinically significant abnormality identified on a medical evaluation
* Male and female volunteers from 18-55 years of age, inclusively, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of: Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea or Child-bearing potential and agrees to use one of the contraception methods listed in the protocol for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point.
* Male subjects must agree to use one of the contraception methods listed in the protocol.
* Nonsmokers defined as abstinence from cigarette smoking for the previous 12 months before enrollment into the study.
* Body mass Index of 19-30 kg/m2.
* FEV1 greater than or equal to 85 percent of the predicted and FEV1/FVC ratio greater than or equal to 0.7 at screening.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

* The subject has a positive pre-study urine drug/ alcohol screen.
* Significant pulmonary disease, such as chronic obstructive pulmonary disease, asthma, or other pulmonary diseases that may affect the pulmonary disposition of study drug or pose a safety risk for oral inhaled study drug.
* Subjects with symptoms of upper respiratory infections at study entry.
* Subjects currently presenting with chronic upper or lower respiratory tract infection, allergic rhinitis, hay fever, or sinusitis.
* Significant psychiatric disease, such as anxiety disorders or psychotic disorders.
* A creatinine clearance less than 70mL/min
* History of regular alcohol consumption within 6 months of the study as defined in the protocol
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer)
* Exposure to more than four experimental medications within 12 months prior to the first dosing day.
* Ingestion of alcohol, grapefruit juice or grapefruit products, caffeine-containing food or beverage with 48 hours prior to the first dose of study medication and continuing through study completion.
* Subjects who have donated blood to the extent where participation in the study would result in excess of 500mL blood donated within a 56 day period.
* History of sensitivity to any of the study medications, or components thereof (including lactose) or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation. In addition, if heparin is used during pharmacokinetic sampling, subjects with a history of sensitivity to heparin or heparin-induced thrombocytopenia should not be enrolled.
* Those who, in the opinion of the investigator, have a risk of non-compliance with study procedures.
* Lack of suitability for participation in this study, for any reason, in the opinion of the investigator.
* Subjects who, after training, are unable to use the study related devices.
* The subject's systolic blood pressure is outside the range of 90-140mmHg, or diastolic blood pressure is outside the range of 45-90mmHg or heart rate is outside the range of 50-100bpm for female subjects or 45-100 bpm for male subjects.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2009-10-12 (Actual); Primary Completion 2009-12-07 (Actual); Study Completion 2009-12-07 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability: AEs, Labs, Vitals | Nineteen days

SECONDARY OUTCOMES:
Pharmacokinetic parameters per protocol | Five days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Weller S, Jones LS, Lou Y, Piscitelli S, Peppercorn A, Ng-Cashin J. Safety, tolerability and pharmacokinetics of orally inhaled zanamivir: a randomized study comparing Rotacap/Rotahaler and Rotadisk/Diskhaler in healthy adults. Antivir Ther. 2013;18(6):827-30. doi: 10.3851/IMP2631. Epub 2013 May 21. PMID 23696221
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 113625 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/113625?search=study&search_terms=113625#rs
- Available data/document: Study Protocol: 113625 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 113625 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113625 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113625 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113625 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113625 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113625 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register